CLINICAL TRIAL: NCT04159350
Title: Point-of-care Anorectal Testing to Predict Outcomes With Biofeedback Therapy: Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: American Gastroenterological Association (Other)
Responsible Party: Principal Investigator, Eric.D.Shah, Director, Center for Gastrointestinal Motility, Esophageal and Swallowing Disorders, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: D19162
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectal Expulsion Device (RED) - Feasibility (Experimental): Feasibility Phase.
  Interventions: Device: Rectal Expulsion Device (RED) - Feasibility
- Rectal Expulsion Device (RED) - Validation (Experimental): Validation Phase.
  Interventions: Device: Rectal Expulsion Device (RED) - Validation

INTERVENTIONS:
Device: Rectal Expulsion Device (RED) - Feasibility — After a complete physical exam at bedside including a digital rectal exam, the patient is turned on their side and RED is gently inserted into the rectum. The patient is then given one minute to expel RED while remaining on their side. If the patient is unable to pass RED, the patient transfers to a commode and attempts to expel the device. If the device is not expelled, the device can be safely removed at bedside and the patient diagnosed with a biofeedback-responsive evacuation disorder.
  The RED device is manufactured by Rose Medical (Grand Rapids, MI) under GMP conditions and final assembly is performed by In2Being (Saline, MI). The device contains accepted technologies that are already in use of humans, namely biomedical grade materials.
  Arms: Rectal Expulsion Device (RED) - Feasibility
Device: Rectal Expulsion Device (RED) - Validation — After a complete physical exam at bedside including a digital rectal exam, the patient is turned on their LEFT side and RED is gently inserted into the rectum. The patient then attempts to expel RED while remaining on their side. If the patient is unable to pass RED, the patient transfers to a commode and attempts to expel the device. If the device is not expelled, the device can be safely removed at bedside and the patient diagnosed with a biofeedback-responsive evacuation disorder.
  The RED device is manufactured by Rose Medical (Grand Rapids, MI) under GMP conditions and final assembly is performed by In2Being (Saline, MI). The device contains accepted technologies that are already in use of humans, namely biomedical grade materials.
  Arms: Rectal Expulsion Device (RED) - Validation

SUMMARY:
To prospectively evaluate the clinical utility of baseline anorectal function testing using a point-of-care device in predicting response of chronically constipated patients to physical therapy biofeedback training.

DETAILED DESCRIPTION:
Chronic constipation affects 10-20% of the US population and can impact quality-of-life to a similar degree as congestive heart failure or rheumatoid arthritis. Notably, 700,000 individuals present to the emergency department for constipation each year in the US and $10 billion is spent annually on laxative therapy. For symptomatic chronic constipation refractory to fiber or laxative therapy, clinical practice guidelines recommend physiological testing to identify abnormalities in anorectal function as the next step5. Abnormal anorectal function testing (including anorectal manometry and balloon expulsion testing) suggests an evacuation disorder, the most common of which is dyssynergic defecation or dyssynergia. Identification of patients with an evacuation disorder as a primary driver of constipation is important since therapy can then be targeted.

To enable standardized, accessible chronic constipation testing for general gastroenterologists, the investigators invented an office-based, point-of-care Rectal Expulsion Device (RED). By incorporating RED into a general gastroenterologist's outpatient visit, chronically constipated individuals with abnormal anorectal function can be identified quickly and directly triaged to biofeedback therapy. Thus, RED offers the possibility of disrupting the current treatment paradigm by enabling an initial biomarker based strategy for patients with chronic constipation. Before such a process of care can be realized, there is a critical need for prospective data to determine the best setting for anorectal function testing in the clinical care pathway. The investigators aim to prospectively evaluate the clinical utility of baseline anorectal function testing using RED in identifying chronically constipated patients with evacuation disorders who would benefit from biofeedback therapy.

The investigators will conduct a 12-week clinical trial enrolling individuals with laxative-refractory chronic constipation. All study participants will undergo RED and traditional lab-based testing at baseline, followed by a standardized three-session biofeedback protocol for dyssynergia.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 18-80 with a body mass index of 18 to 40 kg/m2 and a primary ICD-10 diagnosis for constipation (K59*) or referral for constipation.

  * Does the patient meet Rome IV criteria for functional constipation (FC)?
  * Does the patient report that fiber or laxative therapy has been ineffective to treat constipation in a documented treatment trial for at least two weeks prior to screening?
  * Patient is already scheduled for anorectal manometry and physical therapy as part of routine care.
  * The patient must agree to maintain their current dietary fiber intake and osmotic or bulk-forming laxative regimen (if any) throughout the trial
  * The patient must agree to use stimulant laxatives (such as magnesium citrate [Milk of Magnesia], senna or bisacodyl [Dulcolax]) NO MORE THAN two days per week during the trial
  * Patient must be able to participate in physical therapy for biofeedback
  * Individuals must have health insurance coverage to undergo anorectal function testing and biofeedback therapy as part of their non-study routine clinical care

Exclusion Criteria:

* adults unable to consent, individuals who are not yet adults, pregnant women, and prisoners, as they would be unable to reasonably comply with physical therapy within the duration of the study and would thus undergo unnecessary testing.
* Patient must NOT have tried biofeedback therapy or undergone anorectal manometry previously
* Patient must NOT report prior SURGERY involving the colon or rectum (including surgery for anal fissure, rectal prolapse)
* Patient must NOT recent opioid use within 30 days of enrollment
* Patient must NOT report a neurodegenerative condition (i.e. Parkinson's disease, dementia, multiple sclerosis, spinal cord injury) or uncontrolled inflammatory bowel disease
* Patient must NOT have used linaclotide (Linzess), lubiprostone (Amitiza), plecanatide (Trulance), tegaserod (Zelnorm) or prucalopride (Motegrity) within 30 days prior to enrollment. Patients MUST agree not to use these agents during the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Assessing Change of Global Constipation Symptoms at completion of physical therapy | Week 0 and 12
  The Patient Assessment of Constipation-Symptoms (PAC-SYM) questionnaire is a short, easily-completed instrument for assessing global constipation symptoms. A total PAC-SYM score ranges from 0 to 48.

SECONDARY OUTCOMES:
Measure Change in Bowel Movement Frequency at completion of physical therapy | Week 0 and Week 12
  Measure 7-day average of bowel movement frequency (number of complete spontaneous bowel movements per week and number of spontaneous bowel movements per week). This information will be gathered at week 0 and week 12 in order to measure the change.
Measure Change in Bowel Movement Form at completion of physical therapy | Week 0 and Week 12
  Using the Bristol Stool Scale at week 0 and week 12 measure the change in bowel movement form. The scale breaks down bowel movements into seven different categories based on the appearance of the stool. Stool type 1 indicates hard, lumpy stool and stool type 7 indicates watery stool.
Measure Change in Severity of Straining for Bowel Movements at completion of physical therapy | Week 0 and Week 12
  Using the 5-point Likert scale at week 0 and week 12 to measure the severity of straining during bowel movements. Lower scores indicate less straining. Higher scores indicate more straining.
Measure Change in Severity of Abdominal Discomfort for Bowel Movements at completion of physical therapy | Week 0 and Week 12
  Using the 5-point Likert scale at week 0 and week 12 to measure the severity of abdominal discomfort during bowel movements. Lower scores indicate less abdominal discomfort. Higher scores indicate more abdominal discomfort.
Measure Change in Severity of Bloating for Bowel Movements at completion of physical therapy | Week 0 and Week 12
  Using the 5-point Likert scale at week 0 and week 12 to measure the severity of bloating. Lower scores indicate less bloating. Higher scores indicate more bloating.
Measure Change in Severity of Constipation Severity for Bowel Movements at completion of physical therapy | Week 0 and Week 12
  Using the 5-point Likert scale at week 0 and week 12 to measure the severity of straining during bowel movements. Lower scores indicate less severity. Higher scores indicate more severity.
Assess the Level of Treatment Satisfaction | Week 12
  Using the 5-point Likert scale at week 12 to measure the level of treatment satisfaction. Lower scores indicate less satisfaction. Higher scores indicate more satisfaction.

OTHER OUTCOMES:
Assess the General Health Related Quality of Life at completion of physical therapy | Week 0 and 12
  Using the EuroQOL EQ-5D-5L to assess the health related quality of life at week 0 and week 12. The scores can range from 5 - 25, with lower scores indicating better health for the patient that day.
Assess the Constipation-Related Health Related Quality of Life at completion of physical therapy | Week 0 and 12
  Using the disease specific PAC-QOL to assess the health related quality of life at week 0 and week 12. The minimally important difference to define QoL treatment response in constipation trials is a reduction in composite score of at least 1.0.
Assess work productivity | Week 0 and 12
  Using the WPAI:Constipation v2 instrument to assess work productivity at week 0 and 12.
Level of agreement between binary test results of RED and traditional lab-based testing to detect dyssynergia | Week 0 and 12
  Rome IV and the IAWPG consensus protocol enables a diagnosis of dyssynergia based on agreement among lab-based anorectal function tests. The level of agreement between RED and anorectal manometry on anal relaxation during attempted defecation will be assessed on this outcome.
Level of agreement between binary test results of RED and traditional lab-based testing to detect abnormal rectal sensation | Week 0 and 12
  Rome IV and the IAWPG consensus protocol enables a diagnosis of abnormal rectal sensation based on lab-based anorectal manometry. The level of agreement between RED and anorectal manometry on anal relaxation during attempted defecation will be assessed on this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eric D. Shah, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah ED, Pelletier EA, Greeley C, Sieglinger EE, Sanchez JD, Northam KA, Perrone JA, Curley MA, Navas CM, Ostler TL, Burnett Greeley AR, Martinez-Camblor P, Baker JR, Chey WD. Utility of Anorectal Testing to Predict Outcomes With Pelvic Floor Physical Therapy in Chronic Constipation: Pragmatic Trial. Clin Gastroenterol Hepatol. 2023 Apr;21(4):1070-1081. doi: 10.1016/j.cgh.2022.05.014. Epub 2022 May 29. PMID 35640864
- [Derived] Shah ED, Pelletier EA, Greeley C, Sieglinger EE, Sanchez JD, Northam KA, Perrone JA, Curley MA, Navas CM, Ostler TL, Burnett Greeley AR, Martinez-Camblor P, Baker JR, Harris A, Siegel CA, Chey WD. An Office-Based, Point-of-Care Test Predicts Treatment Outcomes With Community-Based Pelvic Floor Physical Therapy in Patients With Chronic Constipation. Clin Gastroenterol Hepatol. 2023 Apr;21(4):1082-1090. doi: 10.1016/j.cgh.2022.03.022. Epub 2022 Mar 24. PMID 35341952